CLINICAL TRIAL: NCT00354224
Title: A Phase II Study of XELOX in Locally Advanced or Metastatic Gastric Cancer
Brief Title: Capecitabine and Oxaliplatin in Treating Patients With Locally Advanced, Unresectable, or Metastatic Stomach Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to low accrual
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUSC-100829; MUSC-OX-33-064; MUSC-HR-11497; CDR0000484638 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Gastric Cancer
Keywords: recurrent gastric cancer; stage III gastric cancer; stage IV gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oxaliplatin + Capecitabine (Experimental): Patients will receive Oxaliplatin 85 mg/m2/d on day 1, given as a 2-hour infusion in 250 mL of dextrose 5% repeated every 2 weeks. Capecitabine will be administered orally at a dose of 850 mg/m2 twice a day.
  Interventions: Drug: capecitabine; Drug: oxaliplatin

INTERVENTIONS:
Drug: capecitabine
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving capecitabine together with oxaliplatin works in treating patients with locally advanced, unresectable, or metastatic stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response proportion in patients with locally advanced, unresectable, or metastatic gastric cancer treated with capecitabine and oxaliplatin.

Secondary

* Determine the tolerability and toxicity of this regimen in these patients.
* Determine the median and progression-free survival of patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-7. Treatment repeats every 14 days in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed gastric cancer

  * Locally advanced, unresectable, or metastatic disease
* Measurable disease, defined as at least 1 lesion that can be accurately measured in ≥ 1 dimension as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study and for 6 months after completion of study treatment
* Able to swallow
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to fluoropyrimidines or platinum chemotherapy agents
* No uncontrolled intercurrent illness including, but not limited to the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior chemotherapy or radiotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* At least 6 months since prior radiotherapy with capecitabine as a radioenhancer
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent chemotherapy
* No concurrent palliative radiotherapy
* No concurrent hormonal therapy except for the following:

  * Steroids for adrenal failure
  * Hormones for nondisease related conditions (e.g., insulin for diabetes)
  * Intermittent use of dexamethasone as an antiemetic
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uzair B. Chaudhary, MD, Study Chair — Medical University of South Carolina; Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxaliplatin + Capecitabine: Patients will receive Oxaliplatin 85 mg/m2/d on day 1, given as a 2-hour infusion in 250 mL of dextrose 5% repeated every 2 weeks. Capecitabine will be administered orally at a dose of 850 mg/m2 twice a day.
  capecitabine
  oxaliplatin
Period: Overall Study
Arm/Group | Oxaliplatin + Capecitabine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin + Capecitabine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rate as Determined by RECIST.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Every 6 weeks through study completion for up to about 18 weeks
Population: this data was not collected.
Arm/Group | Oxaliplatin + Capecitabine
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Adverse Events
Time Frame: From the start of study treatment through study completion for up to about 18 weeks
Measure: Number; unit: Serious Adverse Events
Arm/Group | Oxaliplatin + Capecitabine
Number analyzed (Participants) | 10
Serious Adverse Events | 4

3. Secondary Outcome: Progression-free Survival
Time Frame: Every 6 weeks through study completion for up to about 18 weeks
Population: data was not collected for this endpoint.
Arm/Group | Oxaliplatin + Capecitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the start of study treatment through study completion for up to about 18 weeks
Description: data for non-serious adverse events was not collected.
Arm/Group | Oxaliplatin + Capecitabine
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin + Capecitabine (N=10)
cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
draining abdominal scar (General disorders) | 1 (1)
supraventricular tachycardia (Cardiac disorders) | 1 (1)
angina (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes